CLINICAL TRIAL: NCT01209884
Title: Metabolomics of Aging: Sub-study of the Healthy Elderly Active Longevity (HEAL) Cohort
Brief Title: Metabolomics of Aging: Sub-study of the Healthy Elderly Active Longevity (HEAL) Study
Acronym: Metabolomics
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Scripps Translational Science Institute
Other Study IDs: SIRB# 10-5416
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample will be collected from each subject after informed consent is obtained
  Blood collection
  Approximately 10mL of blood will be collected. The blood will be collected for the purpose of isolating plasma, as follows:
  1 X 10mls Sodium (Na) Heparin tube
  Blood will be drawn by hospital/clinic phlebotomy services, a nurse or a medical assistant. Blood will be collected from each subject one time.
  Once aliquoted, the plasma will be catalogued in a central registry (LIMS database) and then stored. Metabolite extraction and protein precipitation will be performed to remove proteins and extract the maximum number of metabolites. The samples will be maintained at 4 degrees Celcius in the autosampler and then analyzed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Elderly sub-group: Healthy males between the age of 80-85 years old who have not experienced chronic disease during their lifetime.

SUMMARY:
This research is being done to learn more about healthy aging. We hope to learn which bodily processes or functions are important for the elderly to maintain good health. Metabolites (for example, glucose) are small molecules in our bodies that are used in all bodily reactions. Looking at their levels in healthy elderly people may help researchers find out which processes lead some people to get to disease and others to not.

Metabolites are the basic building blocks for people. They are used to construct larger complexes(such as proteins), relay signals from one part of the body to another, and as a source of energy.

While most people have essentially the same types of metabolites, the relative levels of these metabolites vary from one individual to another. These levels reflect the body's state of growth, development, and reproduction. An appropriate balance in metabolites is important to maintaining general health. Conditions like cancer and diabetes result in disrupted levels of metabolites that are associated with changes in bodily functions. Deviations from normal levels of metabolites can be used as a signature for disease. Researchers have discovered that a disruption in unique metabolite levels is associated with human aging. In this study we hope to learn which, if any, of these disruptions are associated with the onset of age-related disease.

DETAILED DESCRIPTION:
The HEAL study criteria includes subjects who are 80 years of age and older who have not experienced a chronic condition. This sub-study will use plasma samples of up to 100 HEAL subjects to compare the metabolomic findings found within this group with existing young and elderly plasma samples that are currently under analysis at the Siuzdak lab.

The aim of this sub-study is to determine if metabolites that are downregulated in elderly relative to young individuals are similarly downregulated in the Wellderly.

Metabolomics is a rapidly emerging field focused on profiling small, naturally occurring (endogenous) molecules collectively known as the "metabolome." Metabolomics offers a significant advantage over other "omics" sciences (e.g., transcriptomics and proteomics) in that metabolites represent the most

downstream end products of cellular reactions and therefore most closely correlate with the phenotype. Thus, by comparative untargeted profiling, metabolomics provides a powerful strategy for understanding changes associated with a unique phenotype at the molecular level.

Untargeted metabolomics denotes the profiling of all low molecular weight biochemicals, including lipids, hormones, saccharides, nucleotides, organic acids, and amino acids that serve as substrates and products in metabolic pathways. The analytes are measured without specifically "targeting" distinct metabolites or molecules. Untargeted metabolomics has the capacity to implicate unanticipated metabolites or pathways associated with a unique phenotype (i.e., advanced age), and thereby provide great insight into cellular mechanisms and pathobiology. In the latter context, the Siuzdak Laboratory has pioneered a new approach for investigating disease known as therapeutic metabolomics in which cellular pathways associated with disease are identified and then perturbed.

ELIGIBILITY:
INCLUSION CRITERIA

1. Age 80 to 85 years
2. Gender: Male
3. Enrolled in the Healthy Elderly (HEAL) study prior to enrollment in this sub-study
4. Eligible for Blood draw
5. Be reliable, cooperative and willing to comply with all protocol-specified procedures.
6. Able to understand and grant informed consent
7. Be healthy or have mild medical conditions that may be associated with the normal aging process, including:

   1. Hypertension, well controlled with no more than 3 medications
   2. Osteoporosis or Osteopenia
   3. Osteoarthritis
   4. Benign Prostatic Hypertrophy
   5. Cataracts, Glaucoma or Macular Degeneration
   6. Dyslipidemia
   7. Hypothyroidism
   8. Pre-Diabetes/Impaired Fasting Glucose (fasting blood glucose 100-126 mg/dL, if known)
   9. Basal or Squamous Cell Carcinoma

Individuals will be excluded if ANY of the following conditions apply:

EXCLUSION CRITERIA

1. Less than 80 years of age or greater than 85 years of age
2. Gender: Female
3. Currently undergoing treatment with any investigational agents or devices within 30 preceding enrollment in this study.
4. Self-reported history or current diagnosis of significant chronic conditions including"

   1. Any Cancer (including polycythemia; excluding basal or squamous cell carcinoma
   2. Coronary Artery Disease, Myocardial Infarction
   3. Stroke or Transient Ischemic Attack (TIA)
   4. Deep Vein Thrombosis or Pulmonary Embolism
   5. Chronis Renal Disease or Hemodialysis
   6. Significant Auto-Immune or Inflammatory conditions such as Rheumatoid Arthritis, Lupus, Crohn's Disease, etc.
   7. Alzheimer's or Parkinson's Disease
   8. Diabetes (Hemoglobin A1C > 6.5% or fasting glucose > 126 mg/dL or is treated with insulin or oral diabetic medication
   9. Aortic or Cerebral Aneurysm
5. Currently taking any of the following medications on a regular basis:

   1. Chemotherapeutic agents (ex. Tamoxifen, Doxorubicin, Mitoxantrone, bleomycin
   2. Anti-platelet or anticoagulant agents, not including Aspirin (ex. Clopidogrel/Plavix, Dipyridamole/Aggrenox/Persantine, Ticlopidine/Ticlid, Warfarin/Coumadin, Plasugrel, etc.)
   3. Cholinesterase inhibitor for Alzheimer's disease (i.e. Donzepril/Aricept)
   4. Insulin or oral diabetic medication
6. Individual has a significant medical condition which, in the investigator's opinion, may interfere with the individual's optimal participation in the study or would potentially confound interpretation of the individual's phenotype.

Ages: 80 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: General outpatient and community population
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Study the metabolomics of the healthy aging | December 2013

CONTACTS AND LOCATIONS:
Overall Officials: Eric E Topol, MD, Principal Investigator — Scripps Translational Science Institute
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States